CLINICAL TRIAL: NCT03998410
Title: Evaluation of the Diagnostic Value of the TPD System in Determining ADHF Causing Acute Dyspnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to the pandemic
Sponsor: Echosense Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: DOP-27
Record Dates: First submitted 2019-06-23; First posted 2019-06-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-06

CONDITIONS: ADHF
Keywords: ADHF Dyspnea ED

STUDY DESIGN:
Intervention Model Description: Recording Doppler US signals over the right wall chest
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Lung Doppler Signals — Recording Doppler ultrasound on the right chest wall

SUMMARY:
The objective of this study is to evaluate Lung Doppler signals (LDS) among patients presenting to the emergency department with acute dyspnea, in order to determine the diagnostic value of this non-invasive method to discriminate ADHF causing dyspnea from any other cause i.e., non-ADHF causes of dyspnea.

DETAILED DESCRIPTION:
Dyspnea (shortness of breath) is a common symptom affecting as many as 25% of patients seen in ambulatory settings. It can be caused by many different underlying conditions, some of which arise acutely and can be life-threatening, making rapid clinical evaluation and targeted diagnostic studies of central importance. A number of disorders cause dyspnea, including acute decompensated heart failure (ADHF), chronic obstructive pulmonary disease (COPD), asthma, pulmonary embolism, pneumonia, metabolic acidosis, neuromuscular weakness, and others. The overlapping clinical presentations of these conditions and comorbid diseases can make the diagnostic evaluation of dyspnea a significant challenge.

Acute heart failure (AHF) is a major cause of serious morbidity and death in the general population and one of the most common medical causes of hospitalization among people aged over 60. Patients presenting to the ED with ADHF must be evaluated and treated rapidly to ensure the best possible outcomes. The diagnosis should be made as soon as possible and therapy initiated. Delayed diagnosis at presentation may also result in patients being inappropriately transferred to non-specialist wards, resulting in longer stays, increased re-admission and poorer outcomes. The key to improving the time to diagnosis depends on the clinical evaluation alongside a readiness to initiate relevant additional tests.

Previous studies showed that the TPD has the potential to differentiate between the cardiac cause of dyspnea and any other cause.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with acute onset dyspnea (defined as shortness of breath (SOB) at rest or on exertion) and diagnostic uncertainty of etiology where heart failure is in consideration.
* Patients designated to undergo chest X-ray as part of standard of care assessment.

Exclusion Criteria:

* Obvious trauma contributing to dyspnea
* Inability to provide written informed consent
* Not speaking English or Spanish
* Right-sided lobectomy
* Patients with implanted ventricular assist device
* Patient is unable to undergo the TPD test
* Patient is already enrolled in a clinical study with experimental medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of diagnosis | Average of 1 year
  overall accuracy of the TPD system for the determination of ADHF causing acute dyspnea in an ED setting versus the gold standard (GS) diagnosis as determined by the final adjudicated diagnosis

SECONDARY OUTCOMES:
Sensitivity, Specificity, PPV, NPV of TPD diagnosis | Average of 1 year
  Calculate the analysis success parameters

CONTACTS AND LOCATIONS:
Overall Officials: Judd Hollander, MD, Principal Investigator — judd.hollander@jefferson.edu
Locations (3):
- United States (3):
  - Wayne State University, Detroit, Michigan
  - The university of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No